CLINICAL TRIAL: NCT07210593
Title: STrong Relationships to Improve DiabEtes (STRIDE) Pilot
Brief Title: STrong Relationships to Improve DiabEtes Pilot
Acronym: STRIDE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, McKenzie Roddy, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 250845; K23DK140531 (NIH)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; SMART
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Step 1: Optimal First Line Treatment (Experimental): Persons with diabetes (PWD) participants will first be randomized to an optimal first line treatment in order to compare FAMS vs. PEER. PWD participants assigned to Step 1 treatment "FAMS" will have the option to co-enroll a friend/family member as a support person (SP) to receive text message support tailored to the goal set by the linked PWD. PWD participants assigned to Step 1 treatment "PEER" will be paired with another participant to provide each other peer support.
  Interventions: Behavioral: FAMS; Behavioral: PEER
- Experimental: Step 2: Optimal Second Line Treatment (Experimental): All PWD participants will be randomized at month 3 to FAMS or PEER. PWD participants assigned to Step 2 treatment "FAMS" will have the option to co-enroll a friend/family member as a support person (SP) to receive text message support tailored to the goal set by the linked PWD if not previously enrolled. PWD participants assigned to Step 2 treatment "PEER" will be paired with another participant to provide each other peer support. If they had previously enrolled a SP, the SP participant will stop receiving text messages.
  Interventions: Behavioral: FAMS; Behavioral: PEER

INTERVENTIONS:
Behavioral: FAMS — PWD participants will receive FAMS components (monthly phone coaching and text message support for goals and medication adherence) for 3 months. PWD participants will receive high-quality print materials upon enrollment.
  Co-enrolled SP participants will receive high-quality print materials upon enrollment and receive text message support tailored to the goal set by the linked PWD.
Behavioral: PEER — PWD participants will receive PEER components (monthly phone coaching and text message support for goals and medication adherence) for 3 months. PWD participants will receive high-quality print materials upon enrollment PWD participants assigned to PEER will be matched with another PWD participant assigned to peer to provide peer support to each other.

SUMMARY:
This is a pilot and feasibility study for a mobile phone-delivered intervention, called STRIDE (STrong Relationships to Improve DiabEtes), designed to provide support for adults with type 2 diabetes (improve glycemic management and social support). The goal of the study is to examine the feasibility and acceptability of STRIDE.

ELIGIBILITY:
Inclusion Criteria:

PERSONS WITH DIABETES:

* Speaks and reads in English
* 18-75 years old
* Diagnosed with type 2 diabetes
* Receiving outpatient care from a partnering clinic
* Community-dwelling (e.g., not in a nursing facility)
* Prescribed at least one daily diabetes medication
* Owns a mobile phone
* Elevated diabetes distress or low diabetes self-efficacy
* Willing to invite a close friend or family member to co-participate

SUPPORT PERSONS:

* Speaks and reads in English
* 18 years or older
* Owns a mobile phone

Exclusion Criteria:

PERSONS WITH DIABETES

* Unable to communicate by phone
* Currently pregnant
* Currently undergoing treatment for cancer (e.g., radiation, chemotherapy)
* Diagnosed with end-stage renal disease
* Receiving hospice services
* Diagnosed with congestive heart failure
* Diagnosed with dementia
* Diagnosed with schizophrenia
* Demonstrated an inability to receive and respond to a text
* Does not take medication on his/her own/medication administered by someone else SUPPORT PERSONS
* Demonstrated inability to receive & respond to a text
* Unable to communicate by phone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 6 months post-baseline
  Net Promoter Score with scores ranging 0 to 100 where higher scores (scaled score >0) indicate good acceptability
Feasibility (Recruitment) | baseline
  Number of participants screened/week
Feasibility (Recruitment) | baseline
  Proportion of eligible screens who enroll
Feasibility (Treatment Adherence) | 6 months post-baseline
  Proportion of sessions attended
Feasibility (Treatment Adherence) | 6 months post-baseline
  Proportion of interactive texts with response
Feasibility (Assessment Completion) | 3 and 6 months post-baseline
  Proportion of self-report measures completed

SECONDARY OUTCOMES:
Change in Hemoglobin A1c | Baseline and 3 and 6 months post-baseline
  Hemoglobin A1c assessed by mail-in A1c kits from BioQuintex and/or taken from electronic health record (venipuncture or point-of-care) where higher values indicate worse glycemic management
Change in Diabetes Distress | Baseline and 3 and 6 months post-baseline
  Assessed by the Problem Areas in Diabetes (PAID-5) with scores ranging 0-100 where higher scores indicate more emotional, psychological and social distress related to diabetes management (worse)
Change in Psychosocial Well-being | Baseline and 3 and 6 months post-baseline
  Assessed by the World Health Organization - Five Well-Being Index (WHO-5) with scores ranging 0 to 100 where higher scores indicate more well-being (better)
Change in Social Support for Diabetes | Baseline and 3 and 6 months post-baseline
  Assessed by the Diabetes Support Scale (DSS) with scores ranging 12 to 84 where higher scores indicate more social support for diabetes (better)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials, de-identified individual and aggregate survey, clinical, and laboratory data (including raw and recoded data) and associated study documentation (survey codebook; analytic code used in survey and clinical data analyses; standard citation and unique identifier to facilitate attribution of data use) will be made publicly available through the Open Science Framework (OSF).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After study results are posted on clinical trials (required to occur within 1 year of final data collection), scientific data will be submitted to the Open Science Framework (OSF). Under the current repository policies, data will be preserved and available for the wider research community in perpetuity.
Access Criteria: Survey, clinical, and laboratory data and associated study documentation (survey codebook; analytic code used in survey and clinical data analyses; standard citation and unique identifier to facilitate attribution of data use) will be shared and made publicly available through OSF as open access. Survey, clinical, and laboratory data will be made available in csv and text format and will not require the use of specialized tools to be accessed or manipulated. All shared data and documentation will be findable and identifiable using the standard data indexing tools in Open Science Framework.